CLINICAL TRIAL: NCT03259217
Title: Prospects of Clinical Application of Mesenchymal Stem Cells Seeded in Chitosan Scaffold for Diabetic Foot Ulcers
Brief Title: Clinical Application of Mesenchymal Stem Cells Seeded in Chitosan Scaffold for Diabetic Foot Ulcers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Anwar Mohamed Khalifa, DR, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: stem cell in DFU
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Stem Cell Transplant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stem cell product (Experimental): stem cell transplant
  Interventions: Drug: Stem Cell Product

INTERVENTIONS:
Drug: Stem Cell Product — Adipose tissue derived mesenchymal stem cell seeded in Curcumin loaded chitosan nanoparticles into collagen-alginate
  Other Names: mesenchymal stem cells

SUMMARY:
This study will assess the efficacy of application of stem cell in healing of chronic diabetic foot ulcer

DETAILED DESCRIPTION:
Diabetic foot ulcers are a significant and rapidly growing complication of diabetes and its effects on wound healing. Over half of diabetic patients who develop a single ulcer will subsequently develop another ulcer of which the majority will become chronic non-healing ulcers. Over the past decade, the outcomes for patients with ulcers have not improved, despite advances in wound care.These data suggest the importance and necessity of alternative and more effective treatment option for diabetic patients with non-healing ulcers. (Blumberg et al 2012). Stem cell therapy has emerged as a novel therapeutic approach for various diseases including wound repair and tissue regeneration. Mesenchymal stem cells(MSCs) represent an important stem cell population with multipotent capabilities that may have high utility for translational clinical applications. MSCs can differentiate into a variety of cell types, especially fascia originated cells, and provide soluble factors for regeneration of tissues and organs(Şener et al 2015). Adipose tissue is an abundant source of mesenchymal stem cells, which have shown an improved outcome in wound healing studies. Adipose tissue derived stem cells (ASCs )are pluripotent stem cells with the ability to differentiate into different lineages and to secrete paracrine factors initiating tissue regeneration process. The abundant supply of fat tissue, ease of isolation, extensive proliferative capacities ex vivo, and their ability to secrete pro-angiogenic growth factors make them an ideal cell type to use in therapies for the treatment of nonhealing wounds(Hassan et al 2014), However the hostile microenviroment may interfere with viability and efficiency of MSCs injection specially in ischemic tissue , thus increasing needs for new strategies for further improvement of the stem cell therapy of diabetic wounds. Curcumin loaded chitosan nanoparticles into collagen-alginate is a novel biodegradable and biocompatible material that might help a lot in regenerative efficiency in ischemic wound healing

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic patient with diagnosis of neuropathic or neuro-ischemic DFU
2. Chronic non healed diabetic foot ulcer (The wound was determined as non-healing and chronic when the wound was treated with current standard care for diabetic foot ulcer by a wound care specialist for at least 3 months prior to the therapy with less than 40% of wound closure)
3. Strict diabetes control with HbA1c ≤ 7.5%
4. Grade 1 or 2 ulcer on the Wagner scale

Exclusion Criteria:

* 1- Critical ischemia of the target limb, defined by pain at rest and an ankle systolic pressure < 50 mm Hg, or a toe systolic pressure < 30 mm Hg 2- DFU clinically infected as defined by the IDSA/IWGDF criteria, osteomyelitis confirmed by MRI, or other evidence of infection is present 3- Surgery or surgical revascularisation < 2months 4- Collagen tissue diseases , malignant and hematological diseases onset of myocardial infarction or cerebral infarction within the last 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
complete healing | 6 months
  full epithelization of chronic diabetic foot ulcer

SECONDARY OUTCOMES:
Rate of healing | 6 months
  percentage of patients achieving 50 % wound closure
rate of ulcer recurrence | one year
  percentage of patients whose ulcer recurred

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Khalifa, MD, Principal Investigator — lecturer

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sener LT, Albeniz I. Challenge of Mesenchymal Stem Cells Against Diabetic Foot Ulcer. Curr Stem Cell Res Ther. 2015;10(6):530-4. doi: 10.2174/1574888x10666150519092931. PMID 25986622